CLINICAL TRIAL: NCT01849419
Title: Effects of MDMA on Social and Emotional Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 10-120-B; R21DA026570 (NIH)
Record Dates: First submitted 2013-04-23; First posted 2013-05-08 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Drug Addiction
MeSH Terms: conditions — Substance-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group (Experimental): Healthy volunteers received all drug conditions (MDMA, oxytocin, and placebo) using a within-subjects design.
  Interventions: Drug: Within-subjects (MDMA); Drug: Within-subjects (oxytocin); Drug: Within-subjects (placebo)

INTERVENTIONS:
Drug: Within-subjects (MDMA) — This was a within-subjects, double-blind, double-dummy, placebo-controlled experiment during which each participant received a single dose of MDMA (0.75, 1.5 mg/kg) on two session, oxytocin (20 IU) as an active control on one session (see second Intervention), and placebo one session (see third intervention).
Drug: Within-subjects (oxytocin) — This was a within-subjects, double-blind, double-dummy, placebo-controlled experiment during which each participant received oxytocin (20 IU) on one session, MDMA on two sessions (see first Intervention), and placebo on one session (see third Intervention).
Drug: Within-subjects (placebo) — This was a within-subjects, double-blind, double-dummy, placebo-controlled experiment during which each participant received placebo on one session, MDMA on two sessions (see first Intervention), and oxytocin (20 IU) on one session (see second Intervention).

SUMMARY:
The main aim of the study is to investigate the effects of ±3,4-methylenedioxymethamphetamine (MDMA; ecstasy) on social and emotional processing in healthy humans. Ecstasy is a widely used recreational drug, with over 2 million Americans reporting use of the drug in 2006. With this number of users, and evidence that high doses of MDMA are neurotoxic in laboratory animals, the public health implications of ecstasy use may be substantial. Certain subjective effects of this drug distinguish it from other stimulants, and may contribute to its widespread use: That is, users report that ecstasy produces profound feelings of empathy and closeness to others. These so-called 'empathogenic' effects, which may reflect the distinctive neurochemical profile of action of the drug, have yet to be characterized in controlled laboratory studies. The investigators propose to characterize the effects of MDMA on measures of social and emotional processing that may contribute to this 'empathogenic' profile, including measures of emotion recognition, emotional responsiveness and sociability. The investigators will assess effects of MDMA (0, 0.75 and 1.5 mg/kg up to 125 mg) one active control drug (oxytocin: 20 IU) in 100 volunteers who report some prior ecstasy use. Oxytocin will be used because it appears to produce pro-social behavioral effects resembling those attributed to MDMA.

ELIGIBILITY:
Inclusion Criteria:

* 18-35,
* healthy,
* normal weight,
* high school education,
* normal electrocardiogram,
* no psychiatric disorders,
* occasional MDMA use

Exclusion Criteria:

* current medications,
* night shift work,
* abnormal electrocardiogram,
* medical problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: MDMA drug information — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0042542109&QV1=MDMA
- See also: US FDA resources — http://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2010-June 2012, healthy male and non-pregnant female occasional ecstasy users, aged between 18 and 35 years, were recruited through posters, print and internet advertisements and word-of-mouth referrals. All recruitment and study procedures were conducted in a medical laboratory setting.
Pre-assignment Details: Participants were excluded for one of or more of the following reasons: history of adverse effects from ecstasy; current Axis I disorders; medical conditions precluding participation including high blood pressure, abnormal EKG, first degree relatives with heart disease; pregnancy or lactation (females), and significant nasal or sinus condition.
Groups:
- Single Group: Healthy volunteers received all drug conditions/interventions (MDMA, oxytocin, and placebo) using a within-subjects design. Drug order was randomized.
  This was a within-subjects, double-blind, double-dummy, placebo-controlled experiment during which each participant received MDMA (0.75, 1.5 mg/kg), oxytocin (20 IU), and placebo over the course of four experimental sessions. Drug order was randomized for each participant.
Period: Overall Study
Arm/Group | Single Group
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Group: Healthy volunteers received all drug conditions including placebo (within-subjects design).
  Within-subjects (MDMA and placebo): This was a within-subjects, double-blind, double-dummy, placebo-controlled experiment during which each participant received MDMA (0.75, 1.5 mg/kg)and placebo. Participants received oxytocin as an active control on one session (see second Intervention).
  Within-subjects (oxytocin and placebo): This was a within-subjects, double-blind, double-dummy, placebo-controlled experiment during which each participant received oxytocin (20 IU) on one session and placebo on one session. Participants received MDMA on the other two sessions (see first Intervention).
Arm/Group | Single Group
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0
Education [Mean (Standard Deviation); unit: years] | 14.6 (1.4)
MDMA use history [Mean (Standard Deviation); unit: lifetime uses] | 15.0 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Emotional Recognition (MDMA)
Description: Participants complete the Dynamic Emotional Identification Task, or DEIT (Wardle et al. 2012) following MDMA, oxytocin or placebo administration during which they identify emotional facial expressions presented on the screen. Participants completed this task once during each of the sessions.
  In the DEIT, 10 actors performed angry, fearful, sad, and happy expressions, for a total of 40 sequences, which were presented in random order. Each sequence consisted of 50 "frames" progressing from 0 to 100% emotional intensity at 2% steps, producing a color video of an emotional expression developing. Participants were instructed to "press the space bar as soon as you know what expression is being displayed." This ended the sequence and presented options of "angry," "fearful," "sad," and "happy."
  Perception of expressions was quantified as the intensity (0-100 %) of the face when the participant pressed the space bar for correctly identified sequences.
Time Frame: 15 minutes during each session
Measure: Mean (Standard Error); unit: percent intensity
Groups:
- Single Group: Healthy volunteers received all drug conditions/interventions (MDMA, oxytocin, and placebo) using a within-subjects design. Drug order was randomized.
Arm/Group | Single Group
Number analyzed (Participants) | 65
percent intensity | 55.9 (1.5)

2. Primary Outcome: Emotional Recognition (Oxytocin)
Description: Participants completed the Dynamic Emotional Identification Task, or DEIT (Wardle et al. 2012) following MDMA, oxytocin or placebo administration during which they identify emotional facial expressions presented on the screen. Participants completed this task once during each of the sessions.
  In the DEIT, 10 actors performed angry, fearful, sad, and happy expressions, for a total of 40 sequences, which were presented in random order. Each sequence consisted of 50 "frames" progressing from 0 to 100% emotional intensity at 2% steps, producing a color video of an emotional expression developing. Participants were instructed to "press the space bar as soon as you know what expression is being displayed." This ended the sequence and presented options of "angry," "fearful," "sad," and "happy."
  Perception of expressions was quantified as the intensity (0-100 %) of the face when the participant pressed the space bar for correctly identified sequences.
Time Frame: 15 minutes during each session
Measure: Mean (Standard Error); unit: percent intensity
Arm/Group | Single Group
Number analyzed (Participants) | 65
percent intensity | 59.0 (1.4)

3. Primary Outcome: Emotional Recognition (Placebo)
Description: as for outcome 2
Time Frame: 15 minutes during each session
Measure: Mean (Standard Error); unit: percent intensity
Arm/Group | Single Group
Number analyzed (Participants) | 65
percent intensity | 58.9 (1.3)

4. Secondary Outcome: Subjective Response to MDMA (Ratings of 'Feel Drug')
Description: Participants completed this visual analog questionnaire item during which participants selected a rating between 0 ("Not at all") to 100 ("Extremely"). Participants completed this questionnaire item before drug administration and every 30 minutes after drug administration at each session for a total of 6 times. Results are presented as the mean response over the entire session calculated as change from baseline.
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 45.5 (4.5)

5. Secondary Outcome: Subjective Response to Oxytocin (Ratings of 'Feel Drug')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 10.4 (1.5)

6. Secondary Outcome: Subjective Response to Placebo (Ratings of 'Feel Drug')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 10.7 (2.0)

7. Secondary Outcome: Subjective Response to MDMA (Ratings of 'Feel High')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 43.4 (4.4)

8. Secondary Outcome: Subjective Response to Oxytocin (Ratings of 'Feel High')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 10.0 (1.4)

9. Secondary Outcome: Subjective Response to Placebo (Ratings of 'Feel High')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 8.6 (1.8)

10. Secondary Outcome: Subjective Response to MDMA (Ratings of 'Feel Sociable')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 11.7 (3.8)

11. Secondary Outcome: Subjective Response to Oxytocin (Ratings of 'Feel Sociable')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 0.1 (1.5)

12. Secondary Outcome: Subjective Response to Placebo (Ratings of 'Feel Sociable')
Description: as for outcome 4
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | -2.6 (1.9)

13. Secondary Outcome: Cardiovascular Response to MDMA (Heart Rate)
Description: Heart rate (bpm) was assessed before drug administration and repeatedly after drug administration for the each session. Results are presented as the mean response over the entire session calculated as change from baseline.
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Single Group
Number analyzed (Participants) | 65
bpm | 11.1 (2.2)

14. Secondary Outcome: Cardiovascular Response to Oxytocin (Heart Rate)
Description: as for outcome 13
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Single Group
Number analyzed (Participants) | 65
bpm | -4.1 (0.7)

15. Secondary Outcome: Cardiovascular Response to Placebo (Heart Rate)
Description: as for outcome 13
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Single Group
Number analyzed (Participants) | 65
bpm | -4.2 (0.9)

16. Secondary Outcome: Cardiovascular Response to MDMA (Systolic Blood Pressure)
Description: Systolic Blood Pressure (mmHg) was assessed before drug administration and repeatedly after drug administration for the each session. Results are presented as the mean response over the entire session calculated as change from baseline.
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 65
mmHg | 16.4 (1.9)

17. Secondary Outcome: Cardiovascular Response to Oxytocin (Systolic Blood Pressure)
Description: as for outcome 16
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 65
mmHg | 2.8 (0.7)

18. Secondary Outcome: Cardiovascular Response to Placebo (Systolic Blood Pressure)
Description: as for outcome 16
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 65
mmHg | 3.6 (1.1)

19. Secondary Outcome: Cardiovascular Response to MDMA (Diastolic Blood Pressure)
Description: Diastolic Blood Pressure (mmHg) was assessed before drug administration and repeatedly after drug administration for the each session. Results are presented as the mean response over the entire session calculated as change from baseline.
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 65
mmHg | 10.0 (1.5)

20. Secondary Outcome: Cardiovascular Response to Oxytocin (Diastolic Blood Pressure)
Description: as for outcome 19
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 65
mmHg | 2.4 (0.6)

21. Secondary Outcome: Cardiovascular Response to Placebo (Diastolic Blood Pressure)
Description: as for outcome 19
Time Frame: repeatedly during each session
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Single Group
Number analyzed (Participants) | 65
mmHg | 3.1 (0.9)

22. Secondary Outcome: Motivation to Socialize (MDMA)
Description: Participants complete the social choice task following administration of MDMA or placebo during which they choose between spending time 1) talking with another person; 2) sitting quietly alone; or 3) solving word problems. Choices were rated on a scale of 1 to 10 (with 10 indicating the highest level of desire to engage in that activity). The main outcome measure was desire to socialize (i.e., rating of "talking to another person").
Time Frame: 5 minutes during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 5.5 (0.4)

23. Secondary Outcome: Motivation to Socialize (Oxytocin)
Description: as for outcome 22
Time Frame: 5 minutes during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 4.9 (0.3)

24. Secondary Outcome: Motivation to Socialize (Placebo)
Description: as for outcome 22
Time Frame: 5 minutes during each session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 65
units on a scale | 4.6 (0.3)

ADVERSE EVENTS:
Time Frame: Reporting occurred for the full length of the study. But no adverse events occurred.
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

LIMITATIONS AND CAVEATS:
Behavioral measures may not have been obtained at optimal times to detect oxytocin effects. Placebo and oxytocin nasal spray formulations differed slightly. Other potential limitations are the selection of participants, or the doses administered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes